CLINICAL TRIAL: NCT04941495
Title: Effects of Proprioceptive Training in the Management of Chronic Mechanical Neck Pain.
Brief Title: Effects of Cervical Proprioceptive Training in CMNP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mir Arif Hussain (Industry)
Responsible Party: Sponsor-Investigator, Mir Arif Hussain, Director, Aqua Medical Services (Pvt) Ltd
Organization: Aqua Medical Services (Pvt) Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Iqra Raja 00176
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Chronic Neck Pain
Keywords: chronin non traumatic neck pain; Joint position error; Cervical Proprioception; NDI

STUDY DESIGN:
Intervention Model Description: Random allocation will be done through toss coin method into two groups; Conventional Physiotherapy Control group (n=22) and Proprioceptive training Experimental group (n=22).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): It Includes the TENS, Infrared, Isometric and stretching exercises along with the home plan and postural education
  Interventions: Other: conventional physiotherapy
- Experimental Group (Experimental): It Includes the TENS, Infrared, Isometric and stretching exercises along with the home plan and postural education. It also include the cervical proprioceptive training
  Interventions: Other: Cervical proprioceptive training

INTERVENTIONS:
Other: conventional physiotherapy — 1. TENS for 15 minutes on Constant Mode according to patient comfort.
  2. Infrared for 15 minutes.
  3. Isometric exercises: Isometric neck flexion, extension, side bending exercises were given. 3 sets of 10 repetitions each were given. And resistance was given for 6-8 seconds for each movement.
  4. Stretching exercises: Passive stretching for Sternocleidomastoid, short sub occipital muscles, Trapezius & Scalene, Pectoralis Major was given. 3 sets of 10 reps were given and each stretch was maintained for 10 seconds.
  5. Home Plan: self stretches and isometrics.
  6. Postural Education: posture correction in daily life activities in sitting, walking, lying.
  Arms: Control Group
Other: Cervical proprioceptive training — 1. TENS for 15 minutes on Constant Mode according to patient comfort.
  2. Infrared for 15 minutes.
  3. Isometric exercises: Isometric neck flexion, extension, side bending exercises were given. 3 sets of 10 repetitions each were given. And resistance was given for 6-8 seconds for each movement.
  4. Stretching exercises: Passive stretching for Sternocleidomastoid, short sub occipital muscles, Trapezius & Scalene, Pectoralis Major was given. 3 sets of 10 reps were given and each stretch was maintained for 10 seconds.
  5. Home Plan: self stretches and isometrics.
  6. Postural Education: posture correction in daily life activities in sitting, walking, lying.
  7. The patients wearing a cap with a laser pointer attached to it were seated three feet away from the target A, B and C. Start Chart A with a 3 cm, chart B 2cm and chart C 1cm narrow pathway were presented to the patients. The time taken by the patient to complete the pathway without any error was noted.
  Arms: Experimental Group

SUMMARY:
It is a randomized control trial will be conducted at Federal Government Polyclinic hospital on 44 chronic mechanical neck pain patients. Patients will be recruited in the study through non probability purposive sampling. Random allocation will be done through toss coin method into two groups; Conventional Physiotherapy Control group (n=22) and Proprioceptive training Experimental group (n=22). Research data will be collected through structural questionnaires. Tools will be used to collect data are NPRS, NDI, Goniometer (Cervical ROMs) and proprioception.

DETAILED DESCRIPTION:
Neck pain is a very common complaint. In the general population and musculoskeletal practice, it occurs second to low back pain in its frequency. Neck pain has a point prevalence of nearly 13% and lifetime prevalence of nearly 50%. Neck pain and disability are prevalent throughout the industrialized society. It is a common reason for visits in accidents and emergency departments. In Chiropractic treatment, Neck pain is the second most common complaint. It Is the result of fast, mechanical, stressful life, lack of mobility and poor posture. Some injury can also lead to neck pain. Sometimes neck pain lasts for a few days and itself goes away, but when it persists for a long time it results in greater problems. Neck pain is said to be more common in females than in males and in peaks at the middle age. Sedentary lifestyles are contributing to the prevalence of neck pain. Neck pain is one of the most debilitating musculoskeletal problems. Neck problems are a significant source of disability to patients, but they have not been studied in detail as low back pain problems.

Neck pain can be categorized in many ways i.e. Duration(Acute, Sub acute, Chronic), Intensity, Severity, Type(Mechanical, Neuropathic etc.). Among them duration proves to be the best predictor of outcome. Short duration pain have better prognosis than long standing pain. Mechanical Neck Pain is defined as widespread cervical and/or shoulder pain possessing mechanical properties, such as symptoms aggravated by prolonged or abnormal neck posture, neck mobility and/or by palpation of the neck musculature Mechanical pain originates from the spine or by its supporting structures, such as muscles and ligaments. Pain arising from the facet joints eg, arthritis, diskogenic pain, and myofascial pain can be named as Mechanical pain. It is proposed to be associated with several anatomic structures, predominantly facet joints and uncovertebral(Luschka's joints). The risk factors for mechanical neck pain include abnormal posture, stress, substantial lifting and anxiety. Around 15% females and 10% males suffer from Chronic mechanical neck pain at any one time in life. Clinicians find it challenging to prevent a patient from entering into the chronic phase of their condition.

The most mobile part of the vertebral column is the upper cervical spine. And it is at the expense of its mechanical stability. Neuromuscular control to the mobile cervical spine is provided by the highly developed proprioceptive system. Neck pain can lead to disturbed afferent input from the cervical region that may be a possible cause of symptoms such as dizziness, unsteadiness, and visual disturbances. Signs of altered postural stability, cervical proprioception, and head and eye movement control are also said to be the cause of disturbed afferent input.

By an abundance of mechanoreceptors, the proprioceptive system of the cervical spine is very well developed especially from the muscle spindles in the deep segmental upper cervical muscles. Muscle spindle afferent are more important because they are the first ones to operate in proprioception. As compared to the lower cervical spine, the upper cervical spine has an abundance of muscle spindle receptors and greater contributions to reflex activity and connections to the visual and vestibular systems. It concludes that patients with the cause of upper cervical complaints in neck pain have a greater chance for balance and visual disturbances than those with complaints of lower cervical spine.

The ability to maintain body orientation and posture in relation to the surrounding environment is a key process required for normal functions such as coordinated movements. Sensorimotor control of stable upright posture and head and eye movement depends on afferent information from the vestibular, visual and proprioceptive systems, which all together merge in several areas of the Central Nervous System. Proprioception is important for well-adapted sensorimotor control. Proprioception fulfills roles in feedback sensorimotor control and regulation of muscle stiffness, being specifically important for movement acuity, joint stability, coordination, and balance. For head-eye co-ordination and movement control, cervical proprioception is uniquely important. Musculoskeletal disorders due to pain, effusion, trauma, and fatigue alter the normal proprioceptive mechanism.

Neck pain patients are said to have a poor awareness of their head and neck posture, and a few patients are reported to complain about "whopping head" which might be the cause of altered cervical position sense. The rehabilitation procedures in the field of musculoskeletal diseases aim to improve muscular force, joint mobility, and proprioceptive sensibility. Currently, only strength and mobility are evaluated in cervical spine rehabilitation programs, although a wealth of cephalic and neck receptors suggests a major emphasis on proprioceptive information in postural and dynamic functions of the head-neck system.

A study by J Arami and colleagues (2014) on the "Applicability of proprioceptive and endurance measurement protocols to treat patient with chronic non-specific neck pain" was conducted. Chronic neck pain patients were divided into two groups, one of them received endurance training and the other group received proprioceptive training. This study suggested that endurance exercise was a more efficient method for improving endurance and Proprioceptive training was better in resolving joint position error and Pain. Both protocol appeared to be useful in treating patients with chronic non specific neck pain.

Cervicogenic headache is getting common in young adults along with proprioception deficit in the cervical region. In this study, 30 participants of Cervicogenic headache were included. The control group received stretching exercises. The experimental group in addition to stretching received cervical stabilization exercises. Headache disability index and neck proprioception were evaluated before and after the treatment programs. At the end of 4rth week, Headache disability index scores and neck pain and proprioception error improved more in the experimental group. Hence the study concluded that Cervical stabilization exercises along with stretching are more effective in improving neck proprioception and Headache disability index than stretching alone.

The presence of strong coupling between gaze orientation and muscle neck activity has been well documented in humans. This co-ordination between neck motor functions and eye strongly suggest that eye head coupling based rehabilitation program are more appropriate to improve neck proprioception and this afterwards aid in reducing pain. A comparison was done between two groups of neck pain patients one of them receiving the traditional physiotherapy protocol for chronic neck pain and the experimental group received an eye head coupling based rehabilitation program modified from Revel et al., in addition to the traditional protocol given to the other group. The results showed a significant reduction in scores of Neck Pain and Disability scale in both groups with a greater decrease in the experimental subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Mechanical neck pain of Chronic duration (Symptoms present form more than 3 months)
2. Limitation of cervical ROM
3. Age 18-55
4. Men and Women

Exclusion Criteria:

1. Sharp purser test positive
2. Vertebral artery insufficiency test positive Neck pain due to:
3. Inflammatory conditions - infections, ankylosing spondylitis, juvenile arthritis, rheumatoid arthritis and polymyalgia rheumatica.
4. Metabolic - osteoporosis, osteomalacia, Paget's disease, gout.
5. Neoplastic - metastases, myeloma, intrathecal tumours.
6. Referred pain as a result of - angina pectoris, aortic aneurysm, pancoast tumour, diaphragmatic pathology, pharyngial pathology
7. Neck injury due to trauma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2021-06-22 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 2 weeks
  The Numeric Pain Rating Scale (NPRS) is a one-dimensional measure of pain intensity in patients. The NPRS is a numeric version of the visual analog scale (VAS) in which patient selects a number (0-10) from a horizontal line that best depict the intensity of their pain. 0 represents no pain and 10 represents pain as bad as one can imagine.
Neck Disability Index | 2 weeks
  NDI is the most widely used instrument for assessing self rated disability in patients with neck pain. It has a total of 10 sections of the following domain: Pain intensity, personal care, carrying weights, reading, headaches, concentration, work, driving, sleep disturbances and recreational activities.
  Each of the 10 items is scored from 0 (No disability) to 5 (Complete disability).
Range of Motion | 2 weeks
  Range of motion is a movement potential of a joint in which it moves in its possible availble range. For cervical spine active movements of the neck were recorded in sitting postion. Universal goniometer was used to measure patient's active flexion, extension, Left and right side bendings, left and right side rotations.
Cervical Proprioception | 2 weeks
  The treatment protocol used for the patients in experimental group was also used as an outcome measurement tool in this study. Patient's cervical proprioception was measured through a procedure adapted by Clark's Joint position error testing. Patients proprioception was assessed on day one and on the last day of their treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Iqra Raja, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- Federal Government Polyclinic Hospital, Islamabad., Islamabad, Capital, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vernon H, Humphreys K, Hagino C. Chronic mechanical neck pain in adults treated by manual therapy: a systematic review of change scores in randomized clinical trials. J Manipulative Physiol Ther. 2007 Mar-Apr;30(3):215-27. doi: 10.1016/j.jmpt.2007.01.014. PMID 17416276
- [Background] Falla D. Unravelling the complexity of muscle impairment in chronic neck pain. Man Ther. 2004 Aug;9(3):125-33. doi: 10.1016/j.math.2004.05.003. PMID 15245706
- [Background] May S, Gardiner E, Young S, Klaber-Moffett J. Predictor Variables for a Positive Long-Term Functional Outcome in Patients with Acute and Chronic Neck and Back Pain Treated with a McKenzie Approach: A Secondary Analysis. J Man Manip Ther. 2008;16(3):155-60. doi: 10.1179/jmt.2008.16.3.155. PMID 19119405
- [Background] Royuela A, Kovacs FM, Campillo C, Casamitjana M, Muriel A, Abraira V. Predicting outcomes of neuroreflexotherapy in patients with subacute or chronic neck or low back pain. Spine J. 2014 Aug 1;14(8):1588-600. doi: 10.1016/j.spinee.2013.09.039. Epub 2013 Oct 18. PMID 24345468
- [Background] Peterson C, Bolton J, Humphreys BK. Predictors of outcome in neck pain patients undergoing chiropractic care: comparison of acute and chronic patients. Chiropr Man Therap. 2012 Aug 24;20(1):27. doi: 10.1186/2045-709X-20-27. PMID 22920497
- [Background] Fernandez-de-las-Penas C, Palomeque-del-Cerro L, Rodriguez-Blanco C, Gomez-Conesa A, Miangolarra-Page JC. Changes in neck pain and active range of motion after a single thoracic spine manipulation in subjects presenting with mechanical neck pain: a case series. J Manipulative Physiol Ther. 2007 May;30(4):312-20. doi: 10.1016/j.jmpt.2007.03.007. PMID 17509440
- [Background] Kanlayanaphotporn R, Chiradejnant A, Vachalathiti R. The immediate effects of mobilization technique on pain and range of motion in patients presenting with unilateral neck pain: a randomized controlled trial. Arch Phys Med Rehabil. 2009 Feb;90(2):187-92. doi: 10.1016/j.apmr.2008.07.017. PMID 19236972
- [Background] Kristjansson E, Treleaven J. Sensorimotor function and dizziness in neck pain: implications for assessment and management. J Orthop Sports Phys Ther. 2009 May;39(5):364-77. doi: 10.2519/jospt.2009.2834. PMID 19411769
- [Background] Kristjansson E, Leivseth G, Brinckmann P, Frobin W. Increased sagittal plane segmental motion in the lower cervical spine in women with chronic whiplash-associated disorders, grades I-II: a case-control study using a new measurement protocol. Spine (Phila Pa 1976). 2003 Oct 1;28(19):2215-21. doi: 10.1097/01.BRS.0000089525.59684.49. PMID 14520034
- [Background] Rolli Salathe C, Elfering A. A Health- and Resource-Oriented Perspective on NSLBP. ISRN Pain. 2013 Sep 11;2013:640690. doi: 10.1155/2013/640690. eCollection 2013. PMID 27335880
- [Background] Hush JM, Michaleff Z, Maher CG, Refshauge K. Individual, physical and psychological risk factors for neck pain in Australian office workers: a 1-year longitudinal study. Eur Spine J. 2009 Oct;18(10):1532-40. doi: 10.1007/s00586-009-1011-z. Epub 2009 Apr 28. PMID 19399537
- [Background] Descarreaux M, Mayrand N, Raymond J. Neuromuscular control of the head in an isometric force reproduction task: comparison of whiplash subjects and healthy controls. Spine J. 2007 Nov-Dec;7(6):647-53. doi: 10.1016/j.spinee.2006.10.001. Epub 2006 Dec 22. PMID 17509939
- [Background] Clark NC, Roijezon U, Treleaven J. Proprioception in musculoskeletal rehabilitation. Part 2: Clinical assessment and intervention. Man Ther. 2015 Jun;20(3):378-87. doi: 10.1016/j.math.2015.01.009. Epub 2015 Jan 29. PMID 25787919
- [Background] Newcomer KL, Laskowski ER, Yu B, Johnson JC, An KN. Differences in repositioning error among patients with low back pain compared with control subjects. Spine (Phila Pa 1976). 2000 Oct 1;25(19):2488-93. doi: 10.1097/00007632-200010010-00011. PMID 11013501